CLINICAL TRIAL: NCT05893888
Title: Phase 2/3 Run in, Open-Label, Two Arm Study for Safety, Efficacy and Tolerability of PRV111 (Cisplatin Transmucosal System) & PRV211 (Intraoperative Cisplatin System) in Subjects Amenable to Surgery
Brief Title: Safety and Efficacy Study of PRV111 and PRV211 in Subjects With Oral Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Privo Technologies (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-004
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Phase 1/2, Open-Label, Single-Arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pathologically proven and clinically confirmed Tis/CIS of the lip or oral cavity (Experimental): PRV111 Topical Locoregional Delivery Placed Over the Tumor Region Primary Endpoint: Overall Response Rate (ORR) Primary Objective: Demonstrate the safety and efficacy of PRV111 in patients with Carcinoma in Situ (CIS) (WHO 2017)
  Interventions: Drug: PRV111 (Cisplatin Transmucosal System)
- Arm 2: Pathologically proven and clinically confirmed T1-T3, Nx, M0 of the lip or oral cavity (Experimental): Arm 2 PRV211 Intraoperative Locoregional Delivery Placed into the Resected Tumor Bed Primary Endpoint: Safety Primary Objective: Determine Safety of PRV211 in intraoperative setting
  Interventions: Drug: PRV211 (Intraoperative Cisplatin System)

INTERVENTIONS:
Drug: PRV211 (Intraoperative Cisplatin System) — PRV211 system is comprised of two parts, a liquid permeation enhancer (PE) and cisplatin patch. The permeation is brushed onto the resected tumor bed and after 5 minutes the patch can be applied directly over the same area. Apply up to 2 layers of the PRV211 system to the tumor bed post-resection. The duration of the PRV211 treatment takes approximately 10-20 minutes and then the surgeon can continue as planned with the rest of the standard of care procedure. The proposed starting dose is 0.5 mg/cm2 of cisplatin on the tumor bed. This approach can be safe and effective in preventing locoregional recurrence after surgery and eliminating high-risk factors for local recurrence, such as dysplasia at the margins.
  Other Names: Cisplatin
  Arms: Arm 2: Pathologically proven and clinically confirmed T1-T3, Nx, M0 of the lip or oral cavity
Drug: PRV111 (Cisplatin Transmucosal System) — PRV111 (Cisplatin Transmucosal System) is a thin, 2-layer, matrix-type, transmucosal patch consisting of a chitosan matrix layer embedded with cisplatin loaded chitosan particles (CLPs) and a non-woven fabric adhesive unidirectional backing, which is applied to the matrix layer during manufacturing. The patch is self-adhesive. In addition to the PRV111 patch, a separately packaged Permeation Enhancer (PE) Powder for Reconstitution used in conjunction with PRV111. The reconstituted PE Solution is intended to improve the absorption of the cisplatin active ingredient and will be applied prior to patch application.
  Other Names: Cisplatin
  Arms: Arm 1: Pathologically proven and clinically confirmed Tis/CIS of the lip or oral cavity

SUMMARY:
Arm 1 ( Phase 2/3 Run in ):

PRV111: Topical Locoregional Delivery Placed Over the Tumor Region Primary Endpoint: Overall Response Rate (ORR) Primary Objective: Demonstrate the safety and efficacy of PRV111 in patients with Carcinoma in Situ (CIS) (WHO 2017)

Arm 2 (Phase 1) PRV211: Intraoperative Locoregional Delivery Placed into the Resected Tumor Bed Primary Endpoint: Safety Primary Objective: Determine Safety of PRV211 in intraoperative setting

Subject Assignment: Subjects will be assigned to Arm 1 or Arm 2 of this study based on disease staging Arm 1: Pathologically proven and clinically confirmed Tis/CIS of the lip or oral cavity Arm 2: Pathologically proven and clinically confirmed T1-T3, Nx, M0 of the lip or oral cavity

DETAILED DESCRIPTION:
Privo's PRV111 & PRV211 Product Description:

PRV111 (Cisplatin Transmucosal System) is a thin, 2-layer, matrix-type, transmucosal patch consisting of a chitosan matrix layer embedded with cisplatin loaded chitosan particles (CLPs) and a non-woven fabric adhesive unidirectional backing, which is applied to the matrix layer during manufacturing. The patch is self-adhesive.

In addition to the PRV111 patch, a separately packaged Permeation Enhancer (PE) Powder for Reconstitution is used in conjunction with PRV111. The reconstituted PE Solution is intended to improve the absorption of the cisplatin active ingredient and will be applied prior to patch application.

PRV211 is a nanoengineered delivery system intended for intraoperative chemotherapy treatment for all solid tumor surgeries immediately following surgical excision. The goal is to treat the tumor bed locally, eliminating any remaining micrometastases or close margins that are unable to be fully resected while avoiding system circulation.

ARM 1 Study Details PRV111 Topical Treatment

Screening: A screening period of up to 7 days is needed to evaluate subject eligibility for study participation. All subjects will undergo a baseline histopathological assessment at screening (confirming CIS of the oral cavity for inclusion), if an existing diagnosis does not exist. Also at screening, the investigator will determine if the patient requires surgery, and will assess the rest of the inclusion/exclusion criteria to check for eligibility.

Dose limiting Toxicity (DLT): DLT is defined as a clinically significant treatment-emergent AE (TEAE) or laboratory abnormality unrelated to surgery and/or disease progression, concurrent illness, or concomitant therapy within 1-month post-surgery Note: The dosing of 1.5 mg/cm2 per visit in this protocol is comparable to the one used in the prior completed phase 1/2 CLN-001 study, which has shown safety and efficacy causing no dose limiting toxicities (DLTs), related severe adverse events (SAEs) or systemic side effects.

Photo documentation: Tumors will be photographed including anatomic landmarks at each visit, prior to treatment at treatment visits for the ability to compare between visits. Photos are also required for documenting the location of biopsies taken. Additional details are provided in the Lab Manual.

Minimum Required Treatments for Efficacy Assessment: For assessing efficacy, each subject must complete at least 3 treatment visits.

Assessment for Postponement of Surgery: Response Assessment Criteria: If disease is not improved compared to baseline biopsy, subject proceeds to scheduled surgery, otherwise the subject will continue on with the PRV111 treatment regimen.

ARM 2 Study Details PRV211 Intraoperative Treatment

Screening: A screening period of up to 7 days is needed to evaluate subject eligibility for study participation. All subjects will be screened based on the SOC biopsy to obtain baseline histopathology. This biopsy will confirm the stage of the disease to be T1-T3, Nx, M0 of the oral cavity, amenable to surgery. Based on this confirmation, the rest of the inclusion/exclusion criteria will be checked for eligibility.

Safety and Efficacy of PRV211 Treatment: The safety of PRV211 treatment will be determined in the Safety Run-in study described below. Once the safety is determined, a second expansion study can be initiated in another study. The efficacy of PRV211 is determined in the expansion study. This efficacy will be assessed by the incidence of locoregional recurrence at 12 months.

Initial Safety Lead-in Study: This is an open label, safety lead-in phase 1b dose confirmation study in patients with T1-T3, Nx, M0 oral cancer, followed by an expansion phase 2 single arm study as an intraoperative chemotherapy with PRV211. For the purpose of safety detection, if greater than 33% of subjects being evaluated for safety present with dose-limiting toxicities (DLTs), the study is deemed unsafe.

For the Safety Lead-in Study, 3 subjects will be initially enrolled. If more than 1 subject has dose limiting toxicity (DLT), the study stops. Otherwise, 3 additional subjects will be enrolled and if more than 2 DLTs are detected in the total of 6 subjects, the study is deemed unsafe and the study stops. If 2 or less DLTs are observed, the treatment will be considered safe.

At the conclusion of the Safety Lead-in portion (6 patients), if PRV211 is determined to be safe, an expansion study can be initiated. The 6 subjects from the Safety Lead-in study will be included in the expansion study and these patients will be monitored for efficacy.

ELIGIBILITY:
Different diagnosis for ARM 1 & ARM 2, however the rest of inclusion criteria are the same for both arms:

In order to be eligible to participate in the study, an individual must meet all of the following criteria:

• Diagnosis Arm 1: Pathologically proven and clinically confirmed Tis/CIS of the lip or oral cavity Arm 2: Pathologically proven and clinically confirmed T1-T3, Nx,M0 of the lip or oral cavity

Criteria for Inclusion for both ARM 1 & ARM 2:

1. Tumors for which the cytological and architectural changes upon histopathological assessment warrant surgical intervention
2. Adult subjects, men and women, defined by age ≥18 years at the time of screening.
3. Tumor must be accessible, with no evidence of infection or active bleeding.
4. Tumor is amenable to surgical resection within 8 weeks of screening visit (Visit 0).
5. Clinically and/or radiologically measurable tumor.
6. Eastern Collaborative Oncology Group Performance Status of ≤2.
7. Male and female subjects of childbearing potential must agree to use 2 methods of effective contraception from screening and for at least 30 days after the final dose of investigational product. Appropriate birth control is defined as barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine devices, or naturally or surgically sterile (with documentation in the subject's medical records). Postmenopausal women are defined as presenting at least 12 months' natural spontaneous amenorrhea, or at least 6 weeks following surgical menopause (bilateral oophorectomy). Females of childbearing potential must be non-lactating and have a negative serum hCG within 14 days of treatment initiation.
8. Absence of any serious underlying medical conditions which could impair the ability of the subject to participate in the study.
9. Have a life expectancy of ≥3 months.
10. Willing and able to provide written informed consent.
11. Able to return to study site for treatment and follow-up visits as defined in the Protocol.

Criteria for Exclusion for both ARM 1 and ARM 2 (unless specified):

An individual who meets any of the following criteria will be excluded from participation in the study:

1. Subjects that are not eligible for surgery as SOC.
2. Patients with a prior history of invasive squamous cell carcinoma (Arm 1 only)
3. Tumors involving the marginal gingiva (Arm 1 only)
4. Squamous cell carcinoma (SCC) of the oral cavity that received previous radiotherapy.(Arm 1 only)
5. Systemic chemotherapy for the treatment of SCC of the head and neck less than 2 years prior to Screening (Arm 1 only)
6. Concurrent documented malignancy, with the exception of localized SCCs and basal cell carcinoma of the skin Exposure to any investigational agent within 3 months prior to Screening
7. Known allergy or hypersensitivity to platinum-containing agents, or known intolerance to a prior platinum- containing agent, or to any of the excipients, which, in the judgement of the physician will preclude re- exposure to platinum-containing agent
8. Active, uncontrolled infection requiring systemic therapy, such as but not limited to HIV, Syphilis, Hepatitis B, or Hepatitis C
9. Uncontrolled intercurrent illness that would risk subject safety, interfere with the objectives of the Protocol, or limit subject compliance with study requirements, as determined by the Investigator
10. Known or suspected pregnancy, planned pregnancy, or lactation
11. Any medical or psychiatric condition that may compromise the ability to give written informed consent
12. Known diagnosis of oral submucous fibrosis (Arm 1 only)
13. Known diagnosis of trismus (Arm 1 only)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 6-7 months
  Proportion of treated tumors that have a response to PRV111 treatment. Response is defined as either or both: 1) histopathological downgrade of the disease such as partial or complete response as determined by post-treatment biopsies compared to baseline, or 2) clinically measurable tumor volume reduction from baseline of 30% or more from baseline.
Safety assessed via dose-limiting toxicities | 1-month post-surgery and through study completion, ~12-14 months
  Determine a safe dose of PRV211 (Intraoperative Cisplatin System) under the conditions of the trial. For the purpose of safety detection, if greater than 33% of subjects being evaluated for safety present with dose-limiting toxicities (DLTs), the study drug is deemed unsafe.

SECONDARY OUTCOMES:
Event Free Survival | through study completion, ~12-14 months
  An event is defined as: salvage surgery, locoregional recurrence at 12 months or death due to any cause.
Pharmacokinetics: platinum levels in blood | through study completion, ~12-14 months
  whole blood samples will be taken to quantify the amount of cisplatin present.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Miami Cancer Institute, Miami, Florida
  - The University of Chicago, Chicago, Illinois
  - The Cleveland Clinic Foundation, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No